CLINICAL TRIAL: NCT00700154
Title: The Effect of Insulin Infusion on Metabolic Control and Inflammation in Diabetic Patients During Cardio-vascular Intervention and/or Treatment for Acute Foot Ulcer Infection.
Brief Title: Insulin Infusion Diabetes Ulcer
Acronym: IINDU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participants are no longer being examined or receiving intervention
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mats Bonnier, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IICVS_00
Record Dates: First submitted 2008-06-09; First posted 2008-06-18 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus; Insulin Resistance; Hyperglycemia; Surgery; Ulcers; Infection
Keywords: Vascular Surgery; Complications; Hyperglycemia; Insulin infusion; Diabetic ulcers; Infection
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Hyperglycemia; Ulcer; Infections | interventions — Insulin Infusion Systems; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin infusion (aspart) (Experimental)
  Interventions: Procedure: Insulin infusion
- Standard care (No Intervention): Glucose control according to standard care at the ward, i.e., sliding scale insulin at the discretion of responsible physician.

INTERVENTIONS:
Procedure: Insulin infusion — The infusion, a fast acting insulin analog in 1 Unit/ml of NaCl, starts prior the surgery the operation day for all patients and stops during the postoperative care in the control group (conventional therapy), the intervention group continues for three full days with insulin infusion. After the transition day (the fourth day) multiple doses of mixinsulin continues until the study ends 4 weeks after the randomization.
  Other Names: Insulin aspart: NovoRapid
  Arms: Insulin infusion (aspart)

SUMMARY:
Normoglycemia is important for the outcome of surgical and medical conditions. Insulin infusions have been studied to achieve normoglycemia during these circumstances and have proved to be useful. Insulin given by subcutaneous injections has longer duration compared to intravenous given insulin which makes it more difficult to control. The hypothesis behind the trial is the concept that insulin infusion is more effective in reaching normoglycemia in diabetic subjects during treatment for ulcer infections and/or planned cardio-vascular surgery.

* The study evaluates a target controlled insulin infusion or conventional therapy as antidiabetic treatment during ulcer infection and after cardio- vascular surgery.
* Secondary efficacy parameter will be hospital stay, laboratories for inflammation and oxidative stress.

DETAILED DESCRIPTION:
Introduction:

Normoglycemia is important for the outcome of acute surgical and medical conditions. Different insulin infusions have been studied to achieve normoglycemia and have proved to be useful. Insulin given by subcutaneous injections has duration between 3- 36 hours depending on the insulin brand and injection site compared to 10 minutes for intravenous given insulin. Different insulin infusions have been studied to achieve normoglycemia but the biological and chemical effects of insulin infusions have not been studied in routine operative care of patients with diabetes. Therefore, we aim to investigate the importance of normoglycemia for the optimal treatment of ulcer infection and/ or during routine cardio- vascular surgery care among diabetics.

Hypothesis:

Target controlled insulin infusion is more effective in reducing hyperglycemia, improve healing of inflammation and infection in diabetics compared to conventional antidiabetic therapy.

The infusion starts when patients who met the eligibility criteria has signed the informed consent. The intervention group continues for tree full days with insulin infusion. After the transition day (the fourth day) multiple doses of mixinsulin continues until the study ends 4 weeks after the randomization.

Study Design:

This is a randomized prospective, open controlled trial of target controlled insulin infusion vs conventional antidiabetic therapy in diabetic patients. Diabetics planned treated for ulcer infection and/ or after elective cardio- vascular surgery, who met inclusion, not exclusion criteria and choose to participate will be included and randomized.

Duration of study:

The infusion starts when patients who met the eligibility criteria have signed the informed consent and for the surgery group prior the surgery the operation day for all patients and stops during the postoperative care in the control group (conventional therapy). The intervention group continues for three full days with insulin infusion. After the transition day (the fourth day) multiple doses of mixinsulin continues until the study ends 4 weeks after the randomization.

Selection of patients:

Patients with diabetic ulcer infection and/or planned cardio-vascular intervention will be enrolled.

Treatment:

Eligible patients will be randomized to insulin infusion (group 1) for 3 days or therapy according to clinical practise (group 2).

Group 1 (intervention group):

The insulin infusion starts when the patients full fill the eligibility criteria, has signed the informed consent and for the surgery group prior the start of the operation. It controls by regular capillary plasma glucose tests and continues for three days. The infusion stop on the fourth day, the insulin demand is estimated from the last 24 infusion hours by a specific algorithm and divided to 2-4 equal mealtime doses of mixinsulin. The first mealtime dose is given to the breakfast on the fourth day and the infusion continues for another 2 hours where after it is stopped. After the transition day (the fourth day) multiple doses of mixinsulin continues until the study ends 4 weeks after the randomization.

All patients will have a stop visit at the study end.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion if the following criteria are fulfilled:

  * Patients with diabetes type 1 or type 2.
  * Older than 18 years.
  * Patients scheduled for cardio- vascular surgery and/ or acute ulcer infection.
  * Hyperglycaemia: Capillary P-glucose above 8 mmol/L.
  * Informed consent obtained.

Exclusion Criteria:

* Patients having any of the following at randomization will not be included in the study:

  * Unconsciousness: not possible to wake up.
  * Ketoacidosis: pH less or equal to 7.30.
  * Hyperosmolar syndrome: S-Na more or equal to 150 mmol/L.
  * Kidney failure: calculated GFR < 30 mL/min.
  * Pregnancy.
  * Mental condition making the subject unable to understand the concepts and risk of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Plasma glucose levels | 4 weeks

SECONDARY OUTCOMES:
Hospital stay | 4 weeks
HbA1c | 4 weeks
laboratories for inflammation and oxidative stress | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Brismar, Professor, Study Director — Karolinska Institutet; Mats Bonnier, M.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Vascular Surgery, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Malmstedt J, Wahlberg E, Jorneskog G, Swedenborg J. Influence of perioperative blood glucose levels on outcome after infrainguinal bypass surgery in patients with diabetes. Br J Surg. 2006 Nov;93(11):1360-7. doi: 10.1002/bjs.5466. PMID 16779879
- [Background] Bonnier M, Lonnroth P, Gudbjornsdottir S, Attvall S, Jansson PA. Validation of a glucose-insulin-potassium infusion algorithm in hospitalized diabetic patients. J Intern Med. 2003 Feb;253(2):189-93. doi: 10.1046/j.1365-2796.2003.01085.x. PMID 12542559
- [Background] Van den Berghe G, Wilmer A, Milants I, Wouters PJ, Bouckaert B, Bruyninckx F, Bouillon R, Schetz M. Intensive insulin therapy in mixed medical/surgical intensive care units: benefit versus harm. Diabetes. 2006 Nov;55(11):3151-9. doi: 10.2337/db06-0855. PMID 17065355
- [Background] Bastard JP, Maachi M, Lagathu C, Kim MJ, Caron M, Vidal H, Capeau J, Feve B. Recent advances in the relationship between obesity, inflammation, and insulin resistance. Eur Cytokine Netw. 2006 Mar;17(1):4-12. PMID 16613757
- [Background] Brismar K, Fernqvist-Forbes E, Wahren J, Hall K. Effect of insulin on the hepatic production of insulin-like growth factor-binding protein-1 (IGFBP-1), IGFBP-3, and IGF-I in insulin-dependent diabetes. J Clin Endocrinol Metab. 1994 Sep;79(3):872-8. doi: 10.1210/jcem.79.3.7521354.
- [Background] Hadi HA, Suwaidi JA. Endothelial dysfunction in diabetes mellitus. Vasc Health Risk Manag. 2007;3(6):853-76. PMID 18200806
- [Background] Abourizk NN, Vora CK, Verma PK. Inpatient diabetology. The new frontier. J Gen Intern Med. 2004 May;19(5 Pt 1):466-71. doi: 10.1111/j.1525-1497.2004.30133.x. PMID 15109346
- [Background] Collier B, Dossett LA, May AK, Diaz JJ. Glucose control and the inflammatory response. Nutr Clin Pract. 2008 Feb;23(1):3-15. doi: 10.1177/011542650802300103. PMID 18203960
- [Background] Griesdale DE, de Souza RJ, van Dam RM, Heyland DK, Cook DJ, Malhotra A, Dhaliwal R, Henderson WR, Chittock DR, Finfer S, Talmor D. Intensive insulin therapy and mortality among critically ill patients: a meta-analysis including NICE-SUGAR study data. CMAJ. 2009 Apr 14;180(8):821-7. doi: 10.1503/cmaj.090206. Epub 2009 Mar 24. PMID 19318387
- [Background] Sjoholm A, Nystrom T. Inflammation and the etiology of type 2 diabetes. Diabetes Metab Res Rev. 2006 Jan-Feb;22(1):4-10. doi: 10.1002/dmrr.568. PMID 15991254
- [Background] Sjoholm A, Nystrom T. Endothelial inflammation in insulin resistance. Lancet. 2005 Feb 12-18;365(9459):610-2. doi: 10.1016/S0140-6736(05)17912-4. PMID 15708106
- [Background] Campbell RK. Etiology and effect on outcomes of hyperglycemia in hospitalized patients. Am J Health Syst Pharm. 2007 May 15;64(10 Suppl 6):S4-8. doi: 10.2146/ajhp070100. PMID 17494892
- [Background] Van den Berghe G, Schetz M, Vlasselaers D, Hermans G, Wilmer A, Bouillon R, Mesotten D. Clinical review: Intensive insulin therapy in critically ill patients: NICE-SUGAR or Leuven blood glucose target? J Clin Endocrinol Metab. 2009 Sep;94(9):3163-70. doi: 10.1210/jc.2009-0663. Epub 2009 Jun 16. PMID 19531590
- [Background] Kotronen A, Lewitt M, Hall K, Brismar K, Yki-Jarvinen H. Insulin-like growth factor binding protein 1 as a novel specific marker of hepatic insulin sensitivity. J Clin Endocrinol Metab. 2008 Dec;93(12):4867-72. doi: 10.1210/jc.2008-1245. Epub 2008 Sep 16. PMID 18796514
- [Background] King GL. The role of inflammatory cytokines in diabetes and its complications. J Periodontol. 2008 Aug;79(8 Suppl):1527-34. doi: 10.1902/jop.2008.080246. PMID 18673007
- [Background] Pickup JC. Inflammation and activated innate immunity in the pathogenesis of type 2 diabetes. Diabetes Care. 2004 Mar;27(3):813-23. doi: 10.2337/diacare.27.3.813. PMID 14988310
- [Background] Haynes WG. Role of leptin in obesity-related hypertension. Exp Physiol. 2005 Sep;90(5):683-8. doi: 10.1113/expphysiol.2005.031237. Epub 2005 Aug 16. PMID 16105937
- [Background] Gomes F, Telo DF, Souza HP, Nicolau JC, Halpern A, Serrano CV Jr. Obesity and coronary artery disease: role of vascular inflammation. Arq Bras Cardiol. 2010 Feb;94(2):255-61, 273-9, 260-6. doi: 10.1590/s0066-782x2010000200021. English, Portuguese, Spanish. PMID 20428625
- [Background] Arai Y, Kojima T, Takayama M, Hirose N. The metabolic syndrome, IGF-1, and insulin action. Mol Cell Endocrinol. 2009 Feb 5;299(1):124-8. doi: 10.1016/j.mce.2008.07.002. Epub 2008 Jul 11. PMID 18672019
- [Background] Galic S, Oakhill JS, Steinberg GR. Adipose tissue as an endocrine organ. Mol Cell Endocrinol. 2010 Mar 25;316(2):129-39. doi: 10.1016/j.mce.2009.08.018. Epub 2009 Aug 31. PMID 19723556
- [Background] Subramaniam B, Panzica PJ, Novack V, Mahmood F, Matyal R, Mitchell JD, Sundar E, Bose R, Pomposelli F, Kersten JR, Talmor DS. Continuous perioperative insulin infusion decreases major cardiovascular events in patients undergoing vascular surgery: a prospective, randomized trial. Anesthesiology. 2009 May;110(5):970-7. doi: 10.1097/ALN.0b013e3181a1005b. PMID 19387173
- [Background] Van den Berghe G. Endocrine evaluation of patients with critical illness. Endocrinol Metab Clin North Am. 2003 Jun;32(2):385-410. doi: 10.1016/s0889-8529(03)00005-7. PMID 12800538
- [Background] Scurlock C, Raikhelkar J, Mechanick JI. Critique of normoglycemia in intensive care evaluation: survival using glucose algorithm regulation (NICE-SUGAR)--a review of recent literature. Curr Opin Clin Nutr Metab Care. 2010 Mar;13(2):211-4. doi: 10.1097/MCO.0b013e32833571f4. PMID 20010098